CLINICAL TRIAL: NCT00502047
Title: Multicentre, Comparative, Double-Blind, Two-Arm Parallel Clinical Trial of the Effects of Treatment With Plantago Ovata Husk on the Lipid Profile of Patients With Hypercholesterolemia
Brief Title: Effect of the Plantago Ovata Husk on the Lipid Profile of Patients With Hypercholesterolemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rottapharm Spain (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLAN-EC-HIPERL-02; EudraCT number: 2004-002184-24
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2007-07-17 (Estimated); Status verified 2007-07

CONDITIONS: Hypercholesterolemia; Cardiovascular Disease
Keywords: plantago ovata husk; soluble fibre; hypercholesterolemia; cardiovascular risk factor
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Plantago ovata husk

SUMMARY:
The hypothesis of this study is that soluble fibre may contribute to a reduction of the low density lipoprotein cholesterol (LDL-c), and the combined effect with a statin may achieve an optimisation of the cholesterol-lowering effects in adults with several cardiovascular risk factors.

DETAILED DESCRIPTION:
It has been demonstrated that high concentrations of cholesterol and low density lipoprotein cholesterol (LDL, high risk cholesterol) are the major risk factors for heart disease, myocardial infarction and angina pectoris. Moreover, these conditions represent the major cause of death in the Western world.

Of the measures established to reduce blood cholesterol levels, the introduction of consumption of dietary fibre is a novelty. The term dietary fibre defines a variety of substances that are found in plants and are resistant to digestion by human gastrointestinal enzymes.

The studies performed up until now to determine the effects of fibre on blood lipids have demonstrated that consumption of soluble fibre can reduce cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Levels of LDL-c between >130 mg/dl and <189 mg/dl
* Presence at least 1 of the cardiovascular risk factor defined as:
* age above 45 years in men and 55 years in women
* smoker
* high blood pressure
* HDL-c < 40 mg/dl in men and <46 mg/dl in women
* family background of early heart disease
* Patients who have given informed consent
* Patients who will be capable of following diet guidelines

Exclusion Criteria:

* Triglycerides >350 mg/dl
* History of cardiovascular disease

  * treatment with statins prior to the beginning of the trial and who have not dropped out at least 2 months before the beginning of the study
* Diabetes mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2005-09; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To determine the capacity to reduce by 5% the concentrations of plasma LDL-c by treatment with soluble fibre-Plantago ovata husk- added to a low saturated fat diet in patients with moderate hypercholesterolemia. | 16 weeks

SECONDARY OUTCOMES:
To study the combined cholesterol lowering effect of treatment with Plantago ovata husk and statins to achieve the therapeutic objective | 16 weeks
To analyse the effect of Plantago ovata husk fibre on blood pressure | 16 weeks
To evaluate whether the response on plasma lipids is modulated by the polymorphisms of apolipoprotein E, cholesterol ester transfer protein (CETP), apolipoprotein A-V and Fatty acid binding protein 2 (FABP2) | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, MD, phD, Study Chair — Hosp. Universitario San Joan de Reus , Spain; Manuel Castro, MD, phD, Principal Investigator — Hosp. Saint Franciscus Gasthuis, Rotterdam (Netherlands); Eric Brucker, MD, phD, Principal Investigator — Hosp. de la Pitié, Paris (France); Mª Cruz Almaraz, MD, Principal Investigator — Hosp. Universitario Carlos Haya, Málaga (Spain); Xavier Luque, MD, Principal Investigator — Centro de Atención Primaria Alcover, Tarragona (Spain); José Vicente Vaquer, MD, Principal Investigator — Centro de Salud Petrer I, Alicante (Spain); Luis de Teresa, MD, Principal Investigator — Hosp. San Vicente de Raspeig, Alicante (Spain); Silvia Narejos, MD, Principal Investigator — Centro de Atención Primaria Centelles, Barcelona (Spain); Xavier Farrés, MD, Principal Investigator — Centro de Atención Primaria El Remei, Vic, Barcelona (Spain); José Miguel Martínez, MD, Principal Investigator — Centro de Salud Tomás Ortuño, Benidorm, Alicante (Spain)
Locations (1):
- Hosp. Universitario San Joan de Reus, (Spain), Reus, Tarragona, Spain

REFERENCES:
- [Derived] Crescenti A, Sola R, Valls RM, Caimari A, Del Bas JM, Anguera A, Angles N, Arola L. Cocoa Consumption Alters the Global DNA Methylation of Peripheral Leukocytes in Humans with Cardiovascular Disease Risk Factors: A Randomized Controlled Trial. PLoS One. 2013 Jun 26;8(6):e65744. doi: 10.1371/journal.pone.0065744. Print 2013. PMID 23840361